CLINICAL TRIAL: NCT04592666
Title: Almonertinib Plus Pemetrexed and Carboplatin Versus Almonertinib Alone in Advanced NSCLC With EGFR T790M After First- or Second-generation TKIs Therapy: a Randomized, Controlled, Open-label, Phase 2 Study
Brief Title: Almonertinib/Pemetrexed/Carboplatin in EGFR T790M+ Advanced Lung Cancer
Acronym: APPEAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALMO-PEME-CAR-01
Record Dates: First submitted 2020-09-22; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer, Non-small Cell; EGFR T790M; EGFR Gene Mutation
Keywords: lung cancer; EGFR; Combination therapy; Almonertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — aumolertinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combinational therapy (Experimental)
  Interventions: Drug: Almonertinib; Drug: Pemetrexed; Drug: Carboplatin
- Single TKI (Active Comparator)
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — the standard therapy of single agent almonertinib
Drug: Pemetrexed — standard dose
  Arms: Combinational therapy
Drug: Carboplatin — AUC=5
  Arms: Combinational therapy

SUMMARY:
Almonertinib Plus Pemetrexed and Carboplatin Versus Almonertinib Alone in Advanced NSCLC With EGFR T790M After First- or Second-generation TKIs Therapy: a Randomized, Controlled, Open-label, Phase 2 Study

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years old (including 18 and 75 years old);
2. Histologically or cytologically confirmed locally advanced or metastatic (STAGE IIIB-IV) NSCLC does not accept simple sputum smear-based diagnosis;
3. Previous genetic tests confirmed egFR-sensitive mutations, and received one or two generations of EGFR TKI treatment. After drug resistance, it was confirmed to be positive for EGFR T790M mutation by biopsy or free DNA test.
4. The patient has at least one tumor lesion that has not received local treatment such as radiation or biopsy in the screening stage, and can be accurately measured at baseline, with the longest diameter ≥ 10mm at baseline (short diameter ≥ 15mm if lymph nodes are involved).The measurement method chosen is suitable for accurate repeated measurements and can be computed tomography (CT) or magnetic resonance imaging (MRI).If there is only one measurable lesion and no previous local treatment such as irradiation, it can be accepted as the target lesion for baseline evaluation of tumor lesions after at least 14 days of diagnostic biopsy.
5. Life expectancy is at least 3 months;
6. ECOG score: 0-1, with no significant clinical deterioration in the past 2 weeks;
7. The main organs function normally, that is, they meet the following standards:

blood routine examination standards must be in accordance with no blood transfusion and adjuvant therapies (14 days) : A. Hemoglobin (HB) ≥90 g/L; B. Absolute value of neutrophils (ANC) ≥1.5×109/L; C. Platelet (PLT) ≥100×109/L; D. Total bilirubin (TBIL) <1.5 times the upper limit of normal value (ULN); E. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5×ULN, if accompanied by liver metastasis, ALT and AST< 5×ULN; F. Serum Cr<1.25×ULN or endogenous creatinine clearance rate (CCr) > 45 ml/min (Cockcroft-Gault formula);

Exclusion Criteria:

1. Patients who have received three generations of EGFR-TKI treatment;
2. Patients with mixed small cell lung cancer components;
3. Patients with advanced or metastatic disease who have received palliative chemotherapy, or patients with tumor recurrence and metastasis within 6 months after radical surgery with adjuvant chemotherapy;
4. Patients with symptomatic brain metastasis, meningeal metastasis or spinal cord compression;
5. Patients with previous diagnosis of interstitial pneumonia;
6. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite the best medication);
7. with severe cardiovascular disease: Ⅱ magnitude of myocardial ischemia and myocardial infarction, poor control of cardiac arrhythmias (including QTc interphase male 450, female 470 ms or ms or higher);According to NYHA standard, Ⅲ ~ Ⅳ cardiac insufficiency, or heart colour to exceed revealed left ventricular ejection fraction (LVEF) < 50%;
8. abnormal coagulation function (INR >1.5 or prothrombin time (PT) > ULN+4 seconds or APTT > 1.5uln), bleeding tendency or receiving thrombolytic or anticoagulant therapy; Note: Under the condition that the international standard ratio of prothrombin time (INR) ≤1.5, low-dose heparin (daily dosage for adults ranges from 66,000 to 12,000 U) or low-dose aspirin (daily dosage ≤100 mg) is allowed for preventive purposes.
9. Peripheral neuropathy ≥CTCAE 2 is present, except for trauma;
10. Respiratory syndrome (≥CTCAE level 2 dyspnea), uncontrolled serous cavity effusion (including pleural effusion, ascites and pericardial effusion);
11. A wound or fracture that has not been healed for a long time;
12. Severe infections requiring systemic antibiotics;
13. Decompensated diabetes mellitus or other contraindications of high-dose glucocorticoid therapy;
14. Active hepatitis C and/or hepatitis B infection (hepatitis B: HBsAg positive with HBV DNA≥500IU/mL;Hepatitis C: HCV RNA positive);
15. Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
16. Had major surgery or severe traumatic injury, fracture or ulcer within the first 4 weeks;
17. Any contraindications for platinum (carboplatin) and cytotoxic drug (Pemetrexed) treatment;
18. Other conditions deemed inappropriate by the researcher for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2020-10-09 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | from the first cycle of treatment (day one) to two month after the last cycle (each cycle is 21 days)
  progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
based on preliminary results